CLINICAL TRIAL: NCT01621217
Title: Phase I Study of Cetuximab in Combination With 5-fluoruracil, Mitomycin C and Radiotherapy in Patients With Anal Cancer Stage T2 (>4 cm) - T4 N0-3 M0 or Any T N2-3 M0
Acronym: NOAC8
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Lund University Hospital (Other)
Collaborators: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NOAC8.Version1
Record Dates: First submitted 2012-06-14; First posted 2012-06-18 (Estimated); Last update posted 2020-02-28 (Actual); Status verified 2020-02

CONDITIONS: Locally Advanced Cancer in the Anal Region
Keywords: Anal cancer; Locally advanced anal cancer; Cetuximab; 5-fluoruracil; Mitomycin C; Radiotherapy
MeSH Terms: conditions — Anus Neoplasms | interventions — Cetuximab; Mitomycin; Radiotherapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Cetuximab, Mitomycin C, Fluoruracil (Experimental)
  Interventions: Drug: Cetuximab; Drug: Mitomycin C; Drug: 5-Fluoruracil; Radiation: Radiotherapy

INTERVENTIONS:
Drug: Cetuximab — Will be given weekly intravenously during study treatment.
Drug: Mitomycin C — Will be given intravenously twice together with 5-Fluoruracil during study treatment.
Drug: 5-Fluoruracil — Will be given intravenously twice together with Mitomycin C during study treatment
Radiation: Radiotherapy — Radiotherapy, once daily with a total dose of 54 Gy, given in 27 fractions.

SUMMARY:
* To establish maximum tolerated dose of the two cytotoxic drugs 5-fluoruracil and mitomycin C when given together with the antibody cetuximab in patients with locally advanced cancer in the anal region
* To evaluate acute toxicity
* To evaluate late toxicity
* To evaluate response rate
* To evaluate recurrence free survival
* To evaluate overall survival

ELIGIBILITY:
Inclusion Criteria:

* Age over 18 years
* Histologically or cytologically confirmed squamous cell cancer of the anal region (anal canal or anal margin or distal rectum)
* Stage T2 (≥4 cm) - T4 N0-3 M0 or any T N2-3 M0
* ECOG performance status 0-1
* Hb > 100 g/L
* ANC > 1.5 x 10 9/L
* Platelets ≥ 100 x 10 9/L
* Creatinine < 1.5 x ULN
* Bilirubin < 1.5 x ULN
* ALAT < 3.0 x ULN
* Competent to comprehend, sign and date an approved informed consent form

Exclusion Criteria:

* Previous pelvic irradiation
* Previous chemotherapy for anal cancer
* Previous malignancy within the last 5 years, except curatively treated non-melanoma skin cancer or carcinoma in situ of the cervix uteri
* Pregnant or nursing females or patients of child-bearing potential not using adequate methods of birth control
* Patients with active infections or any other serious underlying medical condition, which would impair the ability of the patients to receive the protocol treatment
* Known hypersensitivity to any of the components of the treatment
* Clinically significant cardiovascular disease, e.g. cardiac failure (<12 months before treatment start), unstable angina, congestive heart failure, arrythmia requiring medication, or uncontrolled hypertension
* Known positive test for hepatitis C virus, chronic active hepatitis B infection
* Known HIV infection
* Any other condition or therapy which in the investigator´s opinion may pose a risk to the patient or interfere with the study objectives
* Any investigational agent within 30 days before enrolment
* Surgery (excluding diagnostic biopsy or central venous catheter placement) and/or radiotherapy within 28 days prior to inclusion in the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 21 (Estimated)
Dates: Start 2012-06 (Actual); Primary Completion 2020-01 (Actual); Study Completion 2020-01 (Actual)

PRIMARY OUTCOMES:
To establish maximum tolerable dose of the two cytotoxic drugs 5-fluoruracil and mitomycin C when given together with the antibody cetuximab and radiotherapy in patients with locally advanced cancer in the anal region | Participating patients will be followed during the study period; 8 weeks.

CONTACTS AND LOCATIONS:
Overall Officials: Anders Johnsson, MD, PhD, Principal Investigator — Skåne University Hospital, Dept. of Oncology
Locations (3):
- University Hospital, Dept. of Oncology, Oslo, Norway
- Sweden (2):
  - Skåne University Hospital, Dept. of Oncology, Lund
  - Accademic Hospital, Dept. of Oncology, Uppsala

REFERENCES:
- [Derived] Leon O, Guren MG, Radu C, Gunnlaugsson A, Johnsson A. Phase I study of cetuximab in combination with 5-fluorouracil, mitomycin C and radiotherapy in patients with locally advanced anal cancer. Eur J Cancer. 2015 Dec;51(18):2740-6. doi: 10.1016/j.ejca.2015.08.029. Epub 2015 Nov 18. PMID 26597443